CLINICAL TRIAL: NCT04326920
Title: A Prospective, Randomized, Open-label, Interventional Study to Investigate the Efficacy of Sargramostim (Leukine®) in Improving Oxygenation and Short- and Long-term Outcome of COVID-19 (Corona Virus Disease) Patients With Acute Hypoxic Respiratory Failure.
Brief Title: Sargramostim in Patients With Acute Hypoxic Respiratory Failure Due to COVID-19 (SARPAC)
Acronym: SARPAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Flemish institute of biotechnology (VIB) (Other)
Responsible Party: Principal Investigator, Bart N. Lambrecht, Director, VIB-UGent Center for Inflammation Research, University Hospital, Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARPAC
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: GM-CSF; Acute Lung Injury; Hypoxia; Acute Respiratory Distress Syndrome; Corona virus; COVID-19; SARS (Severe Acute Respiratory Syndrome); Alveolar Macrophage; Acute Hypoxic respiratory failure
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Hypoxia; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active sargramostim treatment group (Active Comparator): Inhaled sargramostim 125mcg twice daily for 5 days on top of standard of care. Upon progression to ARDS and initiation of mechanical ventilator support within the 5 day period, inhaled sargramostim will be replaced by intravenous sargramostim 125mcg/m2 body surface area once daily until the 5 day period is reached. From day 6 onwards, progressive patients in the active group will have the option to receive an additional 5 days of IV sargramostim, based on the treating physician's assessment
  Interventions: Drug: Sargramostim
- Control group (Placebo Comparator): standard of care. Subjects progressing to ARDS and requiring invasive mechanical ventilatory support, from day 6 onwards, will have the option (clinician's decision) to initiate IV sargramostim 125mcg/m2 body surface area once daily for 5 days
  Interventions: Drug: Sargramostim; Other: Control

INTERVENTIONS:
Drug: Sargramostim — Inhalation via mesh nebulizer and/or IV administration upon Clinical deterioration
  Other Names: LEUKINE
Other: Control — Standard of care
  Arms: Control group

SUMMARY:
Phase IV study to evaluate the effectiveness of additional inhaled sargramostim (GM-CSF) versus standard of care on blood oxygenation in patients with COVID-19 coronavirus infection and acute hypoxic respiratory failure.

DETAILED DESCRIPTION:
Leukine® is a yeast-derived recombinant humanized granulocyte-macrophage colony stimulating factor (rhuGM-CSF, sargramostim) and the only FDA approved GM-CSF. GMCSF, a pleiotropic cytokine, is an important leukocyte growth factor known to play a key role in hematopoiesis, effecting the growth and maturation of multiple cell lineages as well as the functional activities of these cells in antigen presentation and cell mediated immunity.

Leukine inhalation or intravenous administration, as an adjuvant therapy, may confer benefit to patients with ARDS (Acute Respiratory Distress Syndrome) due to COVID-19 exposure, who are at significant risk of mortality. While there is no active IND (Investigational New Drug) for Leukine in the proposed patient population, Leukine is being studied in Fase II as an adjuvant therapy in the management of life-threatening infections to boost the hosts innate immune response to fight infection, reduce the risk of secondary infection, and in varied conditions as prevention of infection during critical illness. Inhaled Leukine has also been successfully used as primary therapy to improve oxygenation in patients with disordered gas exchange in the lungs. We propose that based on preclinical and clinical data, Leukine inhalation, as an adjuvant therapy, has an acceptable benefit-risk for use in patients with hypoxic respiratory failure and ARDS due to COVID-19 exposure, who are at significant risk of mortality.

Confirmed COVID19 patients with hypoxic respiratory failure (saturation below 93% on minimal 2 l/min O2) will be randomized to receive sargramostim 125mcg twice daily for 5 days as a nebulized inhalation on top of standard of care, or to receive standard of care treatment. Upon progression of disease requiring initiation of mechanical ventilatory support within the 5 day period, in patients in the active group, inhaled sargramostim will be replaced by intravenous sargramostim 125mcg/m2 body surface area until the 5 day period is reached. From day 6 onwards, progressive patients in the active group will have the option to receive an additional 5 days of IV sargramostim, based on the treating physician's assessment. In the control group progressive disease requiring mechanical ventilatory support, from day 6 onwards, the treating physician will have the option to initiate IV sargramostim 125mcg/m2 body surface area for 5 days. Safety data, including blood leukocyte counts, will be collected in all patients. Efficacy data will also be collected and will include arterial blood gases, oxygenation parameters, need for ventilation, lung compliance, organ function, radiographic changes, ferritin levels, etc. as well as occurrence of secondary bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* Recent (≤2weeks prior to Randomization) confident diagnosis of COVID-19 confirmed by antigen detection and/or PCR (Polymerase Chain Reaction), and/or seroconversion or any other emerging and validated diagnostic test
* In some patients, it may be impossible to get a confident laboratory confirmation of COVID-19 diagnosis after 24h of hospital admission because viral load is low and/or problems with diagnostic sensitivity. In those cases, in absence of an alternative diagnosis, and with highly suspect bilateral ground glass opacities on recent (<24h) chest-CT scan (confirmed by a radiologist and pulmonary physician as probable COVID-19), a patient can be enrolled as probable COVID-19 infected. In all cases, this needs confirmation by later seroconversion.
* Presence of acute hypoxic respiratory failure defined as (either or both)

  * saturation below 93% on minimal 2 l/min O2
  * PaO2/FiO2 below 300
* Admitted to specialized COVID-19 ward
* Age 18-80
* Male or Female
* Willing to provide informed consent

Exclusion Criteria:

* Patients with known history of serious allergic reactions, including anaphylaxis, to human granulocyte-macrophage colony stimulating factor such as sargramostim, yeast-derived products, or any component of the product.
* mechanical ventilation before start of study
* patients with peripheral white blood cell count above 25.000 per microliter and/or active myeloid malignancy
* patients on high dose systemic steroids (> 20 mg methylprednisolone or equivalent)
* patients on lithium carbonate therapy
* Patients enrolled in another investigational drug study
* Pregnant or breastfeeding females (all female subjects regardless of childbearing potential status must have negative pregnancy test at screening)
* Patients with serum ferritin >2000 mcg/ml (which will exclude ongoing HLH)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Lambrecht, Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (4):
  - AZ Sint Jan Brugge, Bruges
  - University Hospital Ghent, Ghent
  - UZ Brussel, Jette
  - AZ Delta Roeselare, Roeselare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosteels C, Van Damme KFA, De Leeuw E, Declercq J, Maes B, Bosteels V, Hoste L, Naesens L, Debeuf N, Deckers J, Cole B, Pardons M, Weiskopf D, Sette A, Weygaerde YV, Malfait T, Vandecasteele SJ, Demedts IK, Slabbynck H, Allard S, Depuydt P, Van Braeckel E, De Clercq J, Martens L, Dupont S, Seurinck R, Vandamme N, Haerynck F, Roychowdhury DF, Vandekerckhove L, Guilliams M, Tavernier SJ, Lambrecht BN. Loss of GM-CSF-dependent instruction of alveolar macrophages in COVID-19 provides a rationale for inhaled GM-CSF treatment. Cell Rep Med. 2022 Dec 20;3(12):100833. doi: 10.1016/j.xcrm.2022.100833. Epub 2022 Nov 15. PMID 36459994
- [Derived] Mehta P, Porter JC, Manson JJ, Isaacs JD, Openshaw PJM, McInnes IB, Summers C, Chambers RC. Therapeutic blockade of granulocyte macrophage colony-stimulating factor in COVID-19-associated hyperinflammation: challenges and opportunities. Lancet Respir Med. 2020 Aug;8(8):822-830. doi: 10.1016/S2213-2600(20)30267-8. Epub 2020 Jun 16. PMID 32559419
- [Derived] Bosteels C, Maes B, Van Damme K, De Leeuw E, Declercq J, Delporte A, Demeyere B, Vermeersch S, Vuylsteke M, Willaert J, Bolle L, Vanbiervliet Y, Decuypere J, Libeer F, Vandecasteele S, Peene I, Lambrecht B. Sargramostim to treat patients with acute hypoxic respiratory failure due to COVID-19 (SARPAC): A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 5;21(1):491. doi: 10.1186/s13063-020-04451-7. PMID 32503663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 87 patients were screened in the period from 25-mar-2020 till 29-sep-2020. 87 patients were included, 81 patients were randomised, 79 patients completed the study
Period: Overall Study
Arm/Group | Active Sargramostim Treatment Group | Control Group
Started | 40 | 41
Completed | 40 | 39
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Sargramostim Treatment Group | Control Group | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 26 | 55
  >=65 years | 11 | 15 | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [46 to 68] | 60 [53 to 69] | 60 [49 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 26 | 25 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 39 | 73
  Black | 4 | 0 | 4
  Arabian | 2 | 2 | 4
Comorbidity at baseline [Count of Participants; unit: Participants]
  Arterial hypertension | 7 | 7 | 14
  Diabetes mellitus | 9 | 7 | 16
  Cardiovascular disease | 0 | 1 | 1
  Chronic kidney disease | 0 | 1 | 1
  Severe liver disease | 0 | 0 | 0
  Chronic lung disease | 0 | 0 | 0
  Cancer | 2 | 2 | 4
  Patients without reported comorbidities | 22 | 23 | 45
Smoking status at baseline [Count of Participants; unit: Participants] — smoking status at baseline
  Participants
    Current | 0 | 3 | 3
    Former | 18 | 16 | 34
    Never | 22 | 22 | 44
Concomitant medication at randomization [Count of Participants; unit: Participants]
  Glucocorticoids | 11 | 9 | 20
  Antiviral drugs (Remdesivir) | 3 | 0 | 3
  Hydroxychloroquine | 24 | 26 | 50
  Antibiotics | 1 | 2 | 3
  Patients without reported concomitant medication | 1 | 4 | 5
6-category ordinal scale at baseline [Count of Participants; unit: Participants] — 6-category ordinal scale at baseline
  Participants
    5 Hospitalized, no supplemental oxygen | 1 | 3 | 4
    4 Hospitalized, supplemental oxygen | 38 | 33 | 71
    3 Hospitalized, Non Invasive Mechanical Ventilation (NIMV) or High Flow Oxygen Device (HFOD) | 1 | 5 | 6
Lab values - C-reactive protein at baseline [Median (Inter-Quartile Range); unit: mg/L] | 73.2 [39.1 to 122.8] | 83 [38.4 to 180] | 74.5 [38.75 to 147.45]
Biomarkers in serum - IL1RA at baseline [Median (Inter-Quartile Range); unit: ng/mL] | 839.3 [595.8 to 1494] | 1288 [905.1 to 2350] | 1162 [678.40 to 1806.00]
Oxygenation - PaO2/FiO2 ratio at baseline [Median (Inter-Quartile Range); unit: ratio] — PaO2/FiO2 ratio is the ratio of the partial pressure of oxygen (PaO2) to the fraction of inspired oxygen (FiO2; PaO2/FiO2).
  ratio | 291.5 [251.5 to 329] | 297 [242 to 319.5] | 295 [248 to 328]
Oxygenation - P(A-a)O2 gradient at baseline [Median (Inter-Quartile Range); unit: mmHg] — partial pressure of oxygen alveolar- arterial ( (P(A-a)O2 gradient)
  mmHg | 50.15 [39.8 to 63.75] | 45.55 [38.6 to 61.75] | 47.65 [38.90 to 61.75]
Lab values - eosinophil count at baseline [Median (Inter-Quartile Range); unit: cells x10^9/L] | 0.01 [0 to 0.1] | 0.02 [0 to 0.09] | 0.02 [0.00 to 0.10]
Lab values - lymphocyte count at baseline [Median (Inter-Quartile Range); unit: cells x10^9/L] | 1.08 [0.83 to 1.4] | 0.88 [0.65 to 1.22] | 1.00 [0.70 to 1.30]
Lab values - ferritin at baseline [Median (Inter-Quartile Range); unit: mcg/L] | 736.5 [446.5 to 1063.5] | 721 [425 to 1068] | 721 [425 to 1068]
Lab values - D-dimer at baseline [Median (Inter-Quartile Range); unit: nmol/L] | 4.36 [3.12 to 5.8] | 3.61 [2.39 to 5.04] | 3.81 [2.79 to 5.31]
Lab values - lactate dehydrogenase at baseline [Median (Inter-Quartile Range); unit: ukat/L] | 4.98 [4.14 to 6.4] | 5.98 [4.31 to 6.86] | 5.26 [4.21 to 6.68]
Lab values - aspartate aminotransferase at baseline [Median (Inter-Quartile Range); unit: ukat/L] | 0.62 [0.44 to 1.01] | 0.65 [0.57 to 0.89] | 0.65 [0.48 to 0.95]
Lab values - alanine aminotransferase at baseline [Median (Inter-Quartile Range); unit: ukat/L] — alanine aminotransferase at baseline
  ukat/L | 0.59 [0.38 to 0.86] | 0.57 [0.4 to 0.92] | 0.58 [0.40 to 0.89]
Lab values - creatinine at baseline [Median (Inter-Quartile Range); unit: micromol/L] | 75.14 [68.07 to 88.4] | 78.68 [68.07 to 92.82] | 77.35 [68.07 to 92.82]
Biomarkers in serum - IL-6 at baseline [Median (Inter-Quartile Range); unit: pg/mL] | 11.47 [4.50 to 21.73] | 11.54 [4.85 to 36.84] | 11.54 [4.85 to 24.90]
Biomarkers in serum - IL-18 at baseline [Median (Inter-Quartile Range); unit: pg/mL] | 101.3 [73.8 to 164.7] | 150.7 [87.13 to 198.3] | 131.00 [80.32 to 184.80]
Biomarkers in serum -C5a at baseline [Median (Inter-Quartile Range); unit: ng/mL] | 11.18 [3.91 to 16.28] | 8.83 [4.52 to 16.06] | 9.94 [4.37 to 16.12]
Biomarkers in serum - GM-CSF at baseline [Median (Inter-Quartile Range); unit: fg/mL] | 9.13 [7.35 to 12.42] | 9.12 [6.82 to 13.39] | 9.12 [7.05 to 12.71]
Biomarkers in serum - TNF at baseline [Median (Inter-Quartile Range); unit: pg/mL] | 16.32 [12.17 to 20.13] | 14.77 [8.53 to 25.91] | 14.99 [10.66 to 22.28]
Body Mass Index (BMI) at baseline [Median (Inter-Quartile Range); unit: kg/m^2] | 28.6 [26 to 33.8] | 27.6 [24.7 to 33.1] | 28.0 [25.0 to 33.4]
Days since symptom onset at baseline [Median (Inter-Quartile Range); unit: day] | 11 [8.5 to 14] | 10 [9 to 13] | 11.0 [9.0 to 13.0]
Days since hospitalization at baseline [Median (Inter-Quartile Range); unit: days] | 3 [2.5 to 4.5] | 3 [3 to 5] | 3.0 [3.0 to 5.0]
Biomarkers in serum - IL-8 at baseline [Median (Inter-Quartile Range); unit: pg/mL] | 22.51 [14.14 to 32.11] | 27.44 [15.91 to 46.49] | 23.99 [15.91 to 39.73]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Oxygenation
Description: Mean Change from Baseline in PaO2/FiO2 on Day 6 or hospital discharge, whichever came first
Time Frame: on Day 6 or hospital discharge, whichever came first
Population: 73 of the 81 patients reached the evaluable primary endpoint. 2 patient discontinued prematurely, 3 patients refused arterial puncture at day 6, 3 patients were excluded because they had a negative P(A-a)O2 gradient at randomization or day 6, signifying an error in FiO2 recording.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 35 | 38
ratio | 25.7 (85.3) | 29.7 (71.88)

2. Secondary Outcome: Mean Change in 6-point Ordinal Scale for Clinical Improvement
Description: The 6-point ordinal scale for clinical improvement is defined as 1 = Death; 2 = Hospitalized, on invasive mechanical ventilation or ECMO (Extracorporeal Membrane Oxygenation) ; 3 = Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4 = Hospitalized, requiring supplemental oxygen; 5 = Hospitalized, not requiring supplemental oxygen; 6 = Not hospitalized. A higher score represent a better outcome
Time Frame: at Baseline, at Day 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
units on a scale | 0.3 (1.0) | 0.3 (1.0)

3. Secondary Outcome: Number of Days in Hospital
Time Frame: through study completion, an average of 5 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
days | 8.5 [6 to 12] | 9.0 [7 to 14]

4. Secondary Outcome: Number of Participants With Nosocomial Infection no./Total no (%)
Time Frame: during hospital admission (up to 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
Participants | 2 | 1

5. Secondary Outcome: Death
Time Frame: at 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
Participants | 2 | 2

6. Secondary Outcome: Number of Participants Progressed to Mechanical Ventilation and/or ARDS
Time Frame: during hospital admission (up to 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
Participants | 7 | 6

7. Secondary Outcome: Time to Clinical Sign Score < 6 for at Least 24h
Description: Clinical Sign score (0-18) by scoring 6 clinical signs from 0 to 3 (0 = absent, 1 = mild, 2 = moderate and 3 = severe): Fever (0 = <37°C; 1 = 37.1-38°C; 2 = 38.1-39°C; 3 = >39°C) last 24h; Cough; Fatigue; Shortness of breath; Diarrhea; Body pain. Higher values represent a worse outcome
Time Frame: During hospital admission (up to 28 days)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
Days | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 6.0]

8. Secondary Outcome: Change in Clinical Sign Score
Description: as for outcome 7
Time Frame: at baseline, at day 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
score on a scale | -2.0 (3.1) | -2.2 (3.0)

9. Secondary Outcome: Change in (National Early Warning Score2) NEWS2 Score
Description: The NEWS2 score standardises the assessment and response to acute illness. Six physiological parameters form the basis of the scoring system:
  respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new confusion, temperature. The total possible score ranges from 0 to 20. The higher the score the greater the clinical risk
Time Frame: at baseline, at day 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
score on a scale | -0.6 (3.1) | -0.4 (3.0)

10. Secondary Outcome: Change in Sequential Organ Failure Assessment (SOFA Score)
Description: The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems (respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems). Score ranges from 0 (best) to 24 (worst) points.
Time Frame: at baseline, at day 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
score on a scale | -0.5 (1.5) | -0.4 (1.2)

11. Secondary Outcome: Change in Ferritin Level
Time Frame: at baseline, at day 6
Measure: Median (95% Confidence Interval); unit: mcg/L
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
mcg/L | -90 [-150 to 34] | -112 [-259 to 118]

12. Secondary Outcome: Change in D-dimer Level
Time Frame: at baseline, at day 6
Measure: Median (95% Confidence Interval); unit: nmol/L
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
nmol/L | -0.71 [-1.79 to 1.33] | -0.44 [-2.90 to 2.46]

13. Secondary Outcome: Change in CRP Level
Time Frame: at baseline, at day 6
Measure: Median (95% Confidence Interval); unit: mg/L
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
mg/L | -43.6 [-69.8 to -21.7] | -43.1 [-73.8 to -22.8]

14. Secondary Outcome: Change in Lymphocyte Count
Time Frame: at baseline, at day 6
Measure: Median (95% Confidence Interval); unit: *cells* x10^9/L
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
*cells* x10^9/L | 0.45 [0.18 to 0.70] | 0.20 [0.02 to 0.56]

15. Secondary Outcome: Change in Eosinophil Count
Time Frame: at baseline, at day 6
Measure: Median (95% Confidence Interval); unit: *cells* x10^9/L
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
*cells* x10^9/L | 0.100 [0.010 to 0.160] | 0.005 [0.000 to 0.073]

16. Secondary Outcome: HRCT (High-Resolution Computed Tomography) Fibrosis Score
Description: The HRCT fibrosis score is a subjective assessment of the overall extent of normal attenuation, reticular abnormalities, honeycombing and traction bronchiectasis . The HRCT findings are graded on a scale of 1-4 based on the classification system: 1. normal attenuation; 2. reticular abnormality; 3. traction bronchiectasis; and 4. honeycombing. The presence of each of the above four HRCT findings is assessed independently in three (upper, middle and lower) zones of each lung. The extent of each HRCT finding was determined by visually estimating the percentage (to the nearest 5%) of parenchymal involvement in each zone. The score for each zone was calculated by multiplying the percentage of the area by the grading scale score (i.e. 1. normal attenuation; 2. reticular abnormality; 3. traction bronchiectasis; and 4. honeycombing). The six zone scores were averaged to determine the total score for each patient. The score ranges from 100 to 400, higher values represent more fibrosis.
Time Frame: at follow-up, 10-20 weeks after day 10 or discharge, whichever comes first
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Sargramostim Treatment Group | Control Group
Number analyzed (Participants) | 40 | 41
score on a scale | 100.8 [100.0 to 102.5] | 102.5 [100.0 to 105.8]

ADVERSE EVENTS:
Time Frame: Timeframe for reporting adverse events: through study completion, an average of 5 months
Arm/Group | Active Sargramostim Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 4/40 | 8/41
Serious Adverse Events (participants affected / at risk) | 6/40 | 6/41
Other Adverse Events (participants affected / at risk) | 22/40 | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Sargramostim Treatment Group (N=40) | Control Group (N=41)
Thormboembolic event (Vascular disorders) | 0 | 1 — pulmonary embolism
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ventilator associated pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspergillus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory deterioration due to underlying MPO-ANCA vasculitis and aspergillosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Increasing hypoxemia due to COVID-19
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 — Progressive symptomatic orthostatism with presyncope
Persistent catatonic state and neurological deficits (Psychiatric disorders) | 1 | 0
Invasive aspergillosis (Infections and infestations) | 1 | 0
Multi-bacterial bacteremia causing hemorrhagic shock (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Sargramostim Treatment Group (N=40) | Control Group (N=41)
Cardiac disorder (Cardiac disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Constipation (Gastrointestinal disorders) | 3 | 6
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Infectious disorder (not COVID-19) (Infections and infestations) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT04326920/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT04326920/SAP_002.pdf